CLINICAL TRIAL: NCT04686409
Title: App-based Symptom Tracking After Corona Vaccination (CoCoV)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Thomas Seufferlein, Professor, Head of Department, University Hospital Ulm
Other Study IDs: CoCoV
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Adverse Events in COVID-19 Vaccination
MeSH Terms: interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: COVID-19 vaccines — Participants will be vaccinated with one of the approved COVID-19 vaccines

SUMMARY:
The study investigates the side effects of different COVID-19 vaccines.

DETAILED DESCRIPTION:
In this observational study side effects of COVID-19 vaccines will be documented using an open-source mobile application. Participants are invited to answer a questionnaire on a daily basis. Common and unknown events are queried and collected. The primary result of this study will be a descriptive analysis of the collected data.

ELIGIBILITY:
Inclusion Criteria:

* received COVID-19 vaccination
* age ≥ 18 years
* mobile device (iOS or Android)

Exclusion Criteria:

* No knowledge of German or English language
* No written informed consent

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult volunteers (≥ 18 years) who received a COVID-19 vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-11 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related side effects | 4 weeks
  Number of participants with treatment-related side effects as assessed by the toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials (status September 2007)

SECONDARY OUTCOMES:
Distribution and deviation of documented side effects | 4 weeks
  Descriptive statistics for different side effects

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Seufferlein, Prof. Dr., Principal Investigator — University Hospital Ulm
Locations (1):
- Universitätsklinikum Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: Undecided